CLINICAL TRIAL: NCT05039671
Title: Feedback and Outcomes for Clinically Useful Student Services (FOCUSS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000030199; 1K08MH116119-01A1 (NIH)
Record Dates: First submitted 2021-08-26; First posted 2021-09-09 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: School-based Mental Health Treatment Services
Keywords: measurement-based care (MBC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measurement-based care (Experimental): Clinicians will receive a 3-hour interactive MBC training followed by six months of post-training consultation. Training and consultation will include how to collect, score, and use student- and parent-reported progress measures with students and families to inform collaborative progress monitoring and treatment decisions.
  Interventions: Behavioral: Measurement-based care (MBC)

INTERVENTIONS:
Behavioral: Measurement-based care (MBC) — Clinicians will receive a 3-hour interactive MBC training followed by six months of post-training consultation. Training and consultation will include how to collect, score, and use student- and parent-reported progress measures with students and families to inform collaborative progress monitoring and treatment decisions.

SUMMARY:
The purpose of the study is to examine the implementation outcomes (i.e., feasibility, appropriateness, acceptability, and fidelity) of MBC in school-based mental health treatment services. The investigators plan to observe the effectiveness of MBC on student engagement and treatment outcomes as a secondary goal. This pilot implementation-effectiveness trial is designed to inform a future, large-scale trial with more participants.

DETAILED DESCRIPTION:
A clustered, multiple-baseline design will be used to examine the impact of implementation support on clinicians' fidelity, use and ratings of MBC appropriateness, acceptability and fidelity. Approximately 50 school-based mental health (SMH) clinicians will be recruited to participate from up to three school districts. All clinicians will receive the same implementation supports; there is no random assignment to condition. Following an initial control period of at least 1 month, school districts will start receiving implementation supports. During the initial control period, baseline MBC use, attitudes, acceptability, feasibility and appropriateness (per clinician self-report) will be collected, as well as needs assessment data from clinician surveys to inform necessary adjustments to the implementation supports. Baseline engagement and student outcomes will be collected after initial clinician training session. MBC implementation outcomes (i.e., MBC use, attitudes, acceptability, appropriateness, and feasibility), engagement and student outcomes will be collected at 3-month and 6-month follow-up during intervention supports, plus a 9-month follow-up interval. This allows clinicians in the two school districts to be compared to each other and to their own baseline. The primary comparison is pre-post ratings of implementation outcomes for all N=50 clinicians. The secondary comparisons are pre-post ratings of engagement and student outcomes, and between-agency differences.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion in the study, a clinician must meet all of the following criteria:

* Female, male or other gender ≥18 years of age at the time of recruitment.
* Provide school-based individual and/or family mental health treatment in an elementary, middle or high school in a participating school district.
* Hold a professional license or certification in their state to provide mental health treatment OR be supervised by a licensed or certified mental health professional in their state.
* English-speaking.
* Ability to provide informed consent.

Exclusion Criteria:

- Clinicians who do not meet all inclusion criteria are excluded. There are no other exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth H. Connors, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Stamford Public Schools, Stamford, Connecticut
  - West Haven Public Schools, West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No
IPD is not available to other researchers at this time, as this is a pilot study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only clinicians were enrolled. Parents were not enrolled in the study. Clinicians were considered "completed" if they completed at least one baseline, 3-month follow up, 6-month follow up, or 9-month follow up survey.
Groups:
- Measurement-based Care Year 1: Clinicians will receive a 3-hour interactive MBC training followed by six months of post-training consultation. Training and consultation will include how to collect, score, and use student- and parent-reported progress measures with students and families to inform collaborative progress monitoring and treatment decisions.
  Measurement-based care (MBC): Clinicians will receive a 3-hour interactive MBC training followed by six months of post-training consultation. Training and consultation will include how to collect, score, and use student- and parent-reported progress measures with students and families to inform collaborative progress monitoring and treatment decisions.
  Year 1 is for academic school year 2021-2022
- Measurement-based Care Year 2: Clinicians will receive a 3-hour interactive MBC training followed by six months of post-training consultation. Training and consultation will include how to collect, score, and use student- and parent-reported progress measures with students and families to inform collaborative progress monitoring and treatment decisions.
  Measurement-based care (MBC): Clinicians will receive a 3-hour interactive MBC training followed by six months of post-training consultation. Training and consultation will include how to collect, score, and use student- and parent-reported progress measures with students and families to inform collaborative progress monitoring and treatment decisions.
  Year 2 is for academic school year 2022-2023.
Period: Overall Study
Arm/Group | Measurement-based Care Year 1 | Measurement-based Care Year 2
Started | 13 | 79
Completed | 12 | 57
Not Completed | 1 | 22

BASELINE CHARACTERISTICS:
Population: Baseline demographics were only collected from participants that completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Measurement-based Care Year 1 | Measurement-based Care Year 2 | Total
Number analyzed (Participants) | 12 | 57 | 69
Age, Customized [Count of Participants; unit: Participants]
  Age: 21-30 | 2 | 8 | 10
  Age: 31-40 | 5 | 16 | 21
  Age: 41-50 | 3 | 16 | 19
  Age: 51-60 | 2 | 12 | 14
  Age: 61 and over | 0 | 5 | 5
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 12 | 51 | 63
  Gender: Male | 0 | 5 | 5
  Gender: Other | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black or African American | 1 | 3 | 4
  Race/Ethnicity: White or Caucasian | 9 | 40 | 49
  Race/Ethnicity: Hispanic or Latino | 1 | 9 | 10
  Race/Ethnicity: Prefer not to answer | 1 | 2 | 3
  Race/Ethnicity: Asian or Asian American | 0 | 1 | 1
  Race/Ethnicity: Multiple Races | 0 | 1 | 1
  Race/Ethnicity: Missing (Did not respond) | 0 | 1 | 1
Professional Discipline [Count of Participants; unit: Participants]
  School Psychology | 3 | 6 | 9
  Social Work | 7 | 44 | 51
  Professional Counseling | 2 | 1 | 3
  Other | 0 | 1 | 1
  Multiple | 0 | 5 | 5
Highest Degree Earned [Count of Participants; unit: Participants]
  Bachelors | 0 | 1 | 1
  Masters | 12 | 55 | 67
  Doctorate | 0 | 1 | 1
Years in Mental Health [Mean (Full Range); unit: years] — Full range for Years in Mental Health refers to the observed range self-reported by clinician participants. "0" years refers to clinicians being in their very first year working in mental health during the study period.
  years | 11.12 [0 to 29] | 16.43 [0 to 40] | 13.78 [0 to 40]
Years in School [Mean (Full Range); unit: years] — Full range for Years in School refers to the observed range self-reported by clinician participants. "0" years refers to clinicians being in their very first year working in schools during the study period.
  years | 10.21 [1 to 25] | 13.45 [1 to 32] | 11.83 [1 to 32]

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician Acceptability of MBC
Description: Change in clinician-reported Acceptability of Intervention Measure (e.g., a score of 5 = completely agree and is most favorable; possible scores range from 1-5)
Time Frame: Baseline, 3-month follow up, 6-month follow up, 9-month follow up
Population: Not all participants were asked to complete each survey that was administered across the study time period. However, the number analyzed varies based on actual survey completion results, which varies by time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Measurement-based Care Year 1: Measurement-based care (MBC): Clinicians will receive a 3-hour interactive MBC training followed by six months of post-training consultation. Training and consultation will include how to collect, score, and use student- and parent-reported progress measures with students and families to inform collaborative progress monitoring and treatment decisions.
  Year 1 is for academic school year 2021-2022
- Measurement-based Care Year 2: Measurement-based care (MBC): Clinicians will receive a 3-hour interactive MBC training followed by six months of post-training consultation. Training and consultation will include how to collect, score, and use student- and parent-reported progress measures with students and families to inform collaborative progress monitoring and treatment decisions.
  Year 2 is for academic school year 2022-2023.
Arm/Group | Measurement-based Care Year 1 | Measurement-based Care Year 2
Number analyzed (Participants) | 12 | 57
score on a scale
  Baseline: number analyzed (Participants) | 12 | 42
  Baseline | 3.96 (0.65) | 3.52 (0.95)
  3-month: number analyzed (Participants) | 6 | 31
  3-month | 4.54 (0.51) | 3.58 (0.87)
  6-month: number analyzed (Participants) | 7 | 0
  6-month | 4.64 (0.63) |
  9-month: number analyzed (Participants) | 9 | 27
  9-month | 4.56 (0.51) | 3.76 (0.75)

2. Primary Outcome: Change in Clinician Appropriateness of MBC
Description: Change in clinician-reported Intervention Appropriateness Measure (e.g., a score of 5 = completely agree and is most favorable; possible scores range from 1-5)
Time Frame: Baseline, 3-month follow up, 6-month follow up, 9-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Measurement-based Care Year 1 | Measurement-based Care Year 2
Number analyzed (Participants) | 12 | 57
score on a scale
  Baseline: number analyzed (Participants) | 12 | 44
  Baseline | 4.13 (0.79) | 3.64 (0.87)
  3-month: number analyzed (Participants) | 6 | 31
  3-month | 4.50 (0.55) | 3.52 (0.99)
  6-month: number analyzed (Participants) | 7 | 0
  6-month | 4.68 (0.55) |
  9-month: number analyzed (Participants) | 9 | 27
  9-month | 4.47 (0.54) | 3.93 (0.8)

3. Primary Outcome: Change in Clinician Feasibility of MBC
Description: Change in clinician-reported Feasibility of Intervention Measure (e.g., a score of 5 = completely agree and is most favorable; possible scores range from 1-5)
Time Frame: Baseline, post training, 3-month follow up, 6-month follow up, 9-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Measurement-based Care Year 1 | Measurement-based Care Year 2
Number analyzed (Participants) | 12 | 57
score on a scale
  Baseline: number analyzed (Participants) | 12 | 44
  Baseline | 3.92 (0.48) | 3.47 (0.86)
  3-Month: number analyzed (Participants) | 6 | 31
  3-Month | 4.29 (0.66) | 3.45 (0.85)
  6-Month: number analyzed (Participants) | 7 | 0
  6-Month | 4.07 (1.16) |
  9-Month: number analyzed (Participants) | 9 | 27
  9-Month | 4.08 (0.64) | 3.74 (0.68)

4. Primary Outcome: Change in Clinician Fidelity to MBC
Description: Monthly fidelity monitoring of ORS measures entered in the online system as evidence of administration with student or parent respondents. A count of participants meeting the established fidelity threshold of 2 or more ORS measures will be calculated each month. Possible scores range from 0-100%.
Time Frame: 9-month follow up (end of school year; end of study period)
Population: Some participants attrited or opted out before the end of the school year.
Measure: Count of Participants; unit: Participants
Arm/Group | Measurement-based Care Year 1 | Measurement-based Care Year 2
Number analyzed (Participants) | 10 | 31
Participants | 9 | 12

5. Primary Outcome: Change in Clinician Use of MBC
Description: Change in clinician-reported Current Assessment Practice Evaluation - Revised (e.g., a score of 100% across all items is most favorable). Possible scores range from 0-100%.
Time Frame: Baseline, post training, 3-month follow up, 6-month follow up, 9-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Measurement-based Care Year 1 | Measurement-based Care Year 2
Number analyzed (Participants) | 12 | 57
score on a scale
  Baseline: number analyzed (Participants) | 12 | 44
  Baseline | 2.23 (4.52) | 19.60 (17.15)
  3-Month: number analyzed (Participants) | 6 | 32
  3-Month | 24.33 (24.63) | 9.81 (15.37)
  6-Month: number analyzed (Participants) | 7 | 0
  6-Month | 31.59 (37.55) |
  9-Month: number analyzed (Participants) | 9 | 24
  9-Month | 21.29 (23.21) | 11.82 (18.38)

6. Primary Outcome: Change in Clinician Acceptability of the PCOMS
Description: Change in clinician-reported Usage Rating Profile - Assessment (e.g., a score of 6 = strongly agree and is most favorable; possible scores range from 1-6. )
Time Frame: 3-month follow up, 6-month follow up, 9-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Measurement-based Care Year 1 | Measurement-based Care Year 2
Number analyzed (Participants) | 10 | 79
score on a scale
  3-Month: number analyzed (Participants) | 6 | 31
  3-Month | 4.62 (0.51) | 3.69 (0.78)
  6-Month: number analyzed (Participants) | 7 | 0
  6-Month | 4.70 (0.54) |
  9-Month: number analyzed (Participants) | 9 | 25
  9-Month | 4.38 (0.59) | 3.95 (0.70)

7. Primary Outcome: Change in Clinician Attitudes Toward Standardized Assessment
Description: Change in clinician-reported Attitudes toward Standardized Assessment-Monitoring and Feedback Scale (e.g., a score of 5 = strongly agree across is most favorable; possible scores range from 1-5)
Time Frame: Baseline, 3-month follow up, 6-month follow up, 9-month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Measurement-based Care Year 1 | Measurement-based Care Year 2
Number analyzed (Participants) | 12 | 79
score on a scale
  Baseline: number analyzed (Participants) | 12 | 46
  Baseline | 3.65 (0.63) | 3.33 (0.59)
  3-Month: number analyzed (Participants) | 6 | 32
  3-Month | 4.31 (0.38) | 3.36 (0.70)
  6-Month: number analyzed (Participants) | 7 | 0
  6-Month | 4.21 (0.48) |
  9-Month: number analyzed (Participants) | 9 | 27
  9-Month | 3.98 (0.57) | 3.49 (0.65)

8. Secondary Outcome: Change in Child Engagement
Description: Data were not collected due to study design changes during the pandemic, which were approved by the Yale IRB and NIMH.
Time Frame: 3-month follow up, 9-month follow up
Population: Data were not collected due to study design changes during the pandemic, approved by the IRB and funder (NIMH).
Arm/Group | Measurement-based Care
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in Child Functioning
Description: Data were not collected due to study design changes during the pandemic, which were approved by the Yale IRB and NIMH.
Time Frame: 3-month follow up, 9-month follow up
Population: Data were not collected due to study design changes during the pandemic, which were approved by the Yale IRB and NIMH.
Arm/Group | Measurement-based Care
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in Parent Engagement
Description: Data were not collected due to study design changes during the pandemic, which were approved by the Yale IRB and NIMH.
Time Frame: Baseline, 3-month follow up, 6-month follow up, 9-month follow up
Population: Data were not collected due to study design changes during the pandemic, which were approved by the Yale IRB and NIMH.
Arm/Group | Measurement-based Care
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Child Emotional and Behavioral Symptoms
Description: Data were not collected due to study design changes during the pandemic, which were approved by the Yale IRB and NIMH.
Time Frame: Baseline, 3-month follow up, 6-month follow up, 9-month follow up
Population: Data were not collected due to study design changes during the pandemic, which were approved by the Yale IRB and NIMH.
Arm/Group | Measurement-based Care
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately 9 months per participant.
Arm/Group | Measurement-based Care Year 1 | Measurement-based Care Year 2
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/79
Other Adverse Events (participants affected / at risk) | 0/13 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT05039671/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT05039671/ICF_001.pdf